CLINICAL TRIAL: NCT02734095
Title: Determining Predictors of Restenosis. Intravascular Ultrasound in the Treatment of Femoropopliteal Lesions
Brief Title: Determining Predictors of Restenosis in Femoropopliteal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Martin Andreas Geiger, Vascular Surgeon, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 52994416.7.0000.5404
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravascular Ultrasound data (Experimental): Intravascular ultrasound measurements after percutaneous transluminal angioplasty and stenting in the treatment of femoropopliteal lesions.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Intravascular ultrasound measurements after percutaneous transluminal angioplasty and stenting in the treatment of femoropopliteal lesions.

SUMMARY:
A prospective, single-center, real-world study on intravascular ultrasound measurements after percutaneous transluminal angioplasty and stenting in the treatment of femoropopliteal lesions.

DETAILED DESCRIPTION:
Intravascular ultrasound is considered important tool in endovascular procedures of coronary territory. Information such as vessel diameter, stent expansion, residual stenosis, helped in better understanding of the disease, treatment and stent behavior.

However, as a different anatomical territory with major hemodynamic differences, many of these concepts could not be reproduced in the femoropopliteal segment.

The purpose of this study is to correlate data collected by intraoperative intravascular ultrasound after the angioplasty procedure with stent placement in femoropopliteal arterial lesions and patency of this revascularization within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Stenotic (>50%) or occlusive atherosclerotic disease of the femoropopliteal arteries;
* Successful lesion passage passed with conventional mechanical guidewires;
* Symptomatic critical limb ischemia (Rutherford 4, 5, 6);
* Life-expectancy of more than 12 months;
* Tha patient must be willing and able to return to the appropriate follow-up times for the duration of the study;
* Te patient must provide written patient informed consent that is approved by the ethics committee.

Exclusion Criteria:

* Patient refusing treatment;
* The reference segment diameter is not suitable fo available balloon and/or stent design;
* Unsuccessfully treated (>30% residual stenosis) proximal inflow limiting arterial stenosis;
* Previously implanted stent(s) or percutaneous transluminal angioplasty at the same lesion site;
* The patient has a known allergy to heparin, Aspirin or other anticoagulant/antiplatelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies;
* The patent has a history of prior life-threatening contrast media reaction;
* The patient is currently enrolled in another investigational device or drug trial;
* The patient is currently breast-feeding, pregnant or intends to become pregnant;
* The patient is mentally ill or retarded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Plaque Burden Measure | intraoperative
  defined as = (external elastic membrane cross-sectional area - lumen cross-sectional area) ÷ external elastic membrane cross-sectional area
Reference Lumen Measure | intraoperative
  defined as = (proximal reference lumen cross-sectional area + distal reference lumen cross-sectional area) x 0.5
Reference Diameter Measure | intraoperative
  defined as = (proximal reference diameter + distal reference diameter) x 0.5
Stent/reference Diameter Ratio Measure | intraoperative
  defined as = stent diameter ÷ reference diameter
Stent Expansion Ratio Measure | intraoperative
  defined as = minimum stent cross-sectional area ÷ reference lumen cross-sectional area
Radial Stent Symmetry Index Measure | intraoperative
  defined as = minimum ÷ maximum stent diameter at minimum stent cross-sectional area
Axial Stent Symmetry Index Measure | intraoperative
  defined as = minimum ÷ maximum stent cross-sectional area
In Stent Restenosis | 12 months (±30 days)

SECONDARY OUTCOMES:
Technical success | intraoperative
  defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater tha 30% and residual stenosis less than 50% by duplex ultrasound (US) imaging.
Freedom of reintervention at each follow-up | Baseline
  defined as freedom from target lesion revascularization (TLR)
Freedom of reintervention at each follow-up | 1 month (± 7 days)
  defined as freedom from target lesion revascularization (TLR)
Freedom of reintervention at each follow-up | 3 months (±30 days)
  defined as freedom from target lesion revascularization (TLR)
Freedom of reintervention at each follow-up | 6 months (±30 days)
  defined as freedom from target lesion revascularization (TLR)
Freedom of reintervention at each follow-up | 12 months (±30 days)
  defined as freedom from target lesion revascularization (TLR)
Limb-salvage rate | Baseline
  defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot)
Limb-salvage rate | 1 month (± 7 days)
  defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot)
Limb-salvage rate | 3 months (±30 days)
  defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot)
Limb-salvage rate | 6 months (±30 days)
  defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot)
Limb-salvage rate | 12 months (±30 days)
  defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot)
Serious adverse events | Baseline
  defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; result in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.
Serious adverse events | 1 month (± 7 days)
  defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; result in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.
Serious adverse events | 3 months (±30 days)
  defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; result in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.
Serious adverse events | 6 months (±30 days)
  defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; result in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.
Serious adverse events | 12 months (±30 days)
  defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; result in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.
Clinical success at follow-up | Baseline
  defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification.
Clinical success at follow-up | 1 month (± 7 days)
  defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification.
Clinical success at follow-up | 3 months (±30 days)
  defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification.
Clinical success at follow-up | 6 months (±30 days)
  defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification.
Clinical success at follow-up | 12 months (±30 days)
  defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Geiger, MD, Principal Investigator — University of Campinas, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DOTTER CT, JUDKINS MP. TRANSLUMINAL TREATMENT OF ARTERIOSCLEROTIC OBSTRUCTION. DESCRIPTION OF A NEW TECHNIC AND A PRELIMINARY REPORT OF ITS APPLICATION. Circulation. 1964 Nov;30:654-70. doi: 10.1161/01.cir.30.5.654. No abstract available. PMID 14226164
- [Background] Dettinger GB. Defending the military family. Am J Psychiatry. 1979 Jun;136(6):855-6. doi: 10.1176/ajp.136.6.855. No abstract available. PMID 443484
- [Background] Pentecost MJ, Criqui MH, Dorros G, Goldstone J, Johnston KW, Martin EC, Ring EJ, Spies JB. Guidelines for peripheral percutaneous transluminal angioplasty of the abdominal aorta and lower extremity vessels. A statement for health professionals from a special writing group of the Councils on Cardiovascular Radiology, Arteriosclerosis, Cardio-Thoracic and Vascular Surgery, Clinical Cardiology, and Epidemiology and Prevention, the American Heart Association. Circulation. 1994 Jan;89(1):511-31. doi: 10.1161/01.cir.89.1.511. No abstract available. PMID 8281692
- [Background] Martin EC, Katzen BT, Benenati JF, Diethrich EB, Dorros G, Graor RA, Horton KM, Iannone LA, Isner JM, Ramee SR, et al. Multicenter trial of the wallstent in the iliac and femoral arteries. J Vasc Interv Radiol. 1995 Nov-Dec;6(6):843-9. doi: 10.1016/s1051-0443(95)71198-8. PMID 8850658
- [Background] Lammer J, Dake MD, Bleyn J, Katzen BT, Cejna M, Piquet P, Becker GJ, Settlage RA. Peripheral arterial obstruction: prospective study of treatment with a transluminally placed self-expanding stent-graft. International Trial Study Group. Radiology. 2000 Oct;217(1):95-104. doi: 10.1148/radiology.217.1.r00se0595. PMID 11012429
- [Background] Gray BH, Olin JW. Limitations of percutaneous transluminal angioplasty with stenting for femoropopliteal arterial occlusive disease. Semin Vasc Surg. 1997 Mar;10(1):8-16. PMID 9068071
- [Background] Ferreira M, Lanziotti L, Monteiro M, Abuhadba G, Capotorto LF, Nolte L, Fearnot N. Superficial femoral artery recanalization with self-expanding nitinol stents: long-term follow-up results. Eur J Vasc Endovasc Surg. 2007 Dec;34(6):702-8. doi: 10.1016/j.ejvs.2007.07.025. Epub 2007 Oct 24. PMID 17920306
- [Background] Bosiers M, Torsello G, Gissler HM, Ruef J, Muller-Hulsbeck S, Jahnke T, Peeters P, Daenens K, Lammer J, Schroe H, Mathias K, Koppensteiner R, Vermassen F, Scheinert D. Nitinol stent implantation in long superficial femoral artery lesions: 12-month results of the DURABILITY I study. J Endovasc Ther. 2009 Jun;16(3):261-9. doi: 10.1583/08-2676.1. PMID 19642788
- [Background] Laird JR, Jain A, Zeller T, Feldman R, Scheinert D, Popma JJ, Armstrong EJ, Jaff MR; Complete SE Investigators. Nitinol stent implantation in the superficial femoral artery and proximal popliteal artery: twelve-month results from the complete SE multicenter trial. J Endovasc Ther. 2014 Apr;21(2):202-12. doi: 10.1583/13-4548R.1. PMID 24754279